CLINICAL TRIAL: NCT02096172
Title: Urine Toxicology With Pharmacogenomic Interpretation Assay: UTOPIA
Acronym: UTOPIA
Status: Withdrawn | Type: Observational
Sponsor: Renaissance RX (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Other Study IDs: 2013-002
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Urine Toxicology

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the impact of pharmacogenomic aspects of drug metabolism on the measurement of drug and drug metabolites on urine drug testing (UDT).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Pharmacogenomic testing within the last 60 days
* Planned UDT

Exclusion Criteria:

* Subject has chronic renal dysfunction, Chronic Kidney Disease Stage 4 or 5
* Subject has a history of abnormal hepatic function within the last 2 years (INR >1.2 not attributable to anticoagulant medications, AST or ALT >1.5x normal, or suspected cirrhosis)
* Subject has a history of malabsorption (short gut syndrome);
* Subject has a history of any gastric or small bowel surgery;
* Subject is currently hospitalized;
* Subject is currently receiving intravenous medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects who are considered candidates for UDT.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Influence of CYP450 drug metabolism on quantitative UDT | 24 months
  Occurrence of genetically-determined abnormal metabolism of drugs tested with UDT, classified as genetic effects on metabolism (GEM) + for rapid metabolizers, GEM 0 for normal metabolizers, and GEM - for slow metabolizers.

SECONDARY OUTCOMES:
Occurrence of illicit drugs detected on UDT and the GEM classification associated with these medications | 24 months
Non-prescribed drugs detected on UDT and the GEM classification associated with these medications | 24 months
False positive immunoassay results, defined as positive immunoassay concurrent with negative quantitative testing | 24 months
Frequency of target drug regimen changes by the treating physician due to pharmacogenomic test results | 24 months
Frequency of illicit drug changes by the subject due to UDT results, as observed at the time of repeat UDT | 24 months
Frequency of non-prescribed drug changes by the subject due to UDT results, as detected at the time of repeat UDT | 24 months